CLINICAL TRIAL: NCT04435717
Title: Unicenter, Randomized, Open-label Clinical Trial on the Efficacy of Tocilizumab in Modifying the Inflammatory Parameters of Patients With COVID-19
Brief Title: Efficacy of Tocilizumab in Modifying the Inflammatory Parameters of Patients With COVID-19 (COVITOZ-01)
Acronym: COVITOZ-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Jose A Perez Molina, Sponsor, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVITOZ-01
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Patients eligible to be included in the study will be randomized in a 1: 1: 1 ratio to receive:
  * TCZ 8 mg / kg (with a maximum of 800 mg) in single dose + usual treatment
  * TCZ 8 mg / kg in two doses at 0 and 12 hours (with a maximum of 800 mg per dose) + usual treatment
  * Usual / standard care treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TCZ 8 mg / kg one dose (Experimental): TCZ 8 mg / kg (with a maximum of 800 mg) in single dose + usual treatment
  Interventions: Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]_#1
- TCZ 8 mg / kg in two (Experimental): TCZ 8 mg / kg in two doses at 0 and 12 hours (with a maximum of 800 mg per dose) + usual treatment
  Interventions: Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]_#1 (2 doses)
- standard care treatment (No Intervention): Usual / standard care treatment

INTERVENTIONS:
Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]_#1 — Tocilizumab 20 MG/ML Intravenous (one dose)
  Arms: TCZ 8 mg / kg one dose
Drug: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]_#1 (2 doses) — Tocilizumab 20 MG/ML Intravenous ( two doses)
  Other Names: Tocilizumab 20 MG/ML Intravenous Solution [ACTEMRA]_#1
  Arms: TCZ 8 mg / kg in two

SUMMARY:
unicenter, randomized, open-label clinical trial on the efficacy of tocilizumab in modifying the inflammatory parameters of patients with COVID-19.

DETAILED DESCRIPTION:
National, unicenter, randomized, open-label, controlled phase II clinical trial with a drug marketed and administered under conditions of use other than those approved.

The study is designed to evaluate the effect of adding Tocilizumab to standard or standard of care for patients infected with COVID-19 and diagnosed with mild-moderate pneumonia.

78 patients are expected to be included in the study in a single center in Spain. The study includes a selection and randomization period, and a 28-day follow-up period (or until death, or premature withdrawal, whichever is earlier). Once the patients complete the study, they will continue with their usual follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age who have given their informed consent. This will be collected verbally and will be recorded in the medical record by the investigating doctor.
2. The patient is diagnosed with mild-moderate SARS-CoV-2 pneumonia confirmed microbiologically ≤7 days before randomization, and presents:

   to. Basal oxygen saturation> 90% b. CURB-65 ≤1 c. PaO2 / FiO2≥300 or SatO2 / FiO2≥315
3. The patient is hospitalized or meets hospital admission criteria.
4. The patient is not expected to enter the ICU or die in the next 24 hours.

Exclusion Criteria:

1. Participants in another simultaneous clinical trial.
2. Use of other immunomodulators.
3. Coinfection with the hepatitis B virus (detectable AgSup-HBV).
4. Pregnancy (or planning to become pregnant during the course of the study), or lactation period.
5. Presence of laboratory abnormalities of grade ≥ 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in IL-12 values in the 3 study groups from the start of treatment (D0) and on days D + 1 and D + 3. | Day1 and Day3.
  Average increase in IL-12 values in the 3 study groups from the start of treatment (D0) and on days D + 1 and D + 3.

SECONDARY OUTCOMES:
Progression of pneumonia | Day3, Day7 and Day28
  Percentage of patients per group with progression of pneumonia in Day3, Day 7 and Day28
PaO2/FiO2 | Day3, Day7 and Day28
  Proportion of patients with PaO2 / FiO2 <300 (or SatO2 / FiO2 ≤315) at some point in the evolution.
cause mortality to 28 days after started treatment | Day3, Day7 and Day28
  cause mortality to 28 days after started treatment
Length of hospital stay | Day3, Day7 and Day28
  Length of hospital stay
patients requiring Intensive Care Unit admission | Day3, Day7 and Day28
  Percentage of patients requiring Intensive Care Unit admission
evolution of inflammatory parameters IL12 | Day0, Day3 and Day7
  IL-12 levels at Day 7
evolution of inflammatory parameters IL-10, IL-1, IL-6, IL-17 and IFN-gamma | Day0, Day3 and Day7
  IL-10, IL-1, IL-6, IL-17 and IFN-gamma levels on days Day 0, Day1, Day 3 and Day 7
evolution of inflammatory parameters Procalcitonin (PCT), | Day0, Day3 and Day7
  Procalcitonin (PCT), levels on days Day0, Day1, Day3 and Day 7
  * 7
evolution of inflammatory parameters C-reactive protein (PCR), | Day0, Day3 and Day7
  C-reactive protein (PCR),levels on days Day0, Day1, Day3 and Day 7
  * 7
evolution of inflammatory parameters D-dimer | Day0, Day3 and Day7
  D-dimer levels on days Day0, Day1, Day3 and Day 7
  * 7
evolution of inflammatory parameters and ferritin | Day0, Day3 and Day7
  ferritin levels on days Day0, Day1, Day3 and Day 7
  * 7
pharmacokinetics of tocilizumab Cmin | Day0, Day1 Day3 and Day7
  Cmin,on Day0, Day1, Day3 and Day7. On day 0 (D0), blood samples will be collected 12 hours after the infusion of each dose of tocilizumab in both experimental treatment groups.
pharmacokinetics of tocilizumab Cmax | days Day0, Day1 Day3 and Day7
  Cmax,on Day0, Day1, Day3 and Day7. On day 0 (D0), blood samples will be collected 12 hours after the infusion of each dose of tocilizumab in both experimental treatment groups.
pharmacokinetics of tocilizumab Cmedia | days Day0, Day1 Day3 and Day7
  Cmedia,on Day0, Day1, Day3 and Day7. On day 0 (D0), blood samples will be collected 12 hours after the infusion of each dose of tocilizumab in both experimental treatment groups.
pharmacokinetics of tocilizumab Tmax | days Day0, Day1 Day3 and Day7
  Tmax,on Day0, Day1, Day3 and Day7. On day 0 (D0), blood samples will be collected 12 hours after the infusion of each dose of tocilizumab in both experimental treatment groups.
pharmacokinetics of tocilizumab AUC | days Day0, Day1 Day3 and Day7
  AUC,on Day0, Day1, Day3 and Day7. On day 0 (D0), blood samples will be collected 12 hours after the infusion of each dose of tocilizumab in both experimental treatment groups.
Adverse event | days Day0, Day3, Day7 and Day28
  Serious and non-serious adverse events.
Adverse event to cause the treatment interruption. | days Day0, Day3, Day7 and Day28
  Adverse events to cause the treatment interruption.
Adverse event Abnormalities in laboratory | days Day0, Day3, Day7 and Day28
  Abnormalities in laboratory findings unrelated to COVID-19 disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No